CLINICAL TRIAL: NCT06703658
Title: A Phase I, Randomised, Single-blind, Placebo-controlled, Single and Repeated Dose-escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD5004 in Healthy Japanese Participants and With Type 2 Diabetes Mellitus
Brief Title: A Study to Investigate Multiple Ascending Doses of AZD5004 in Healthy Japanese Participants and Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7260C00003
Record Dates: First submitted 2024-10-29; First posted 2024-11-25 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants; Type 2 Diabetes
Keywords: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A-AZD5004 (Experimental): Participants will receive AZD5004 orally.
  Interventions: Drug: AZD5004(Part A)
- Part A-Placebo (Placebo Comparator): Participants will receive matching Placebo orally.
  Interventions: Drug: Placebo(Part A)
- Part B-AZD5004 (Experimental): Participants will receive AZD5004 orally.
  Interventions: Drug: AZD5004(Part B)
- Part B-Placebo (Placebo Comparator): Participants will receive matching Placebo orally.
  Interventions: Drug: Placebo(Part B)

INTERVENTIONS:
Drug: AZD5004(Part A) — Single dose of AZD5004 oral on Day1
  Arms: Part A-AZD5004
Drug: Placebo(Part A) — Single dose of placebo oral on Day1
  Arms: Part A-Placebo
Drug: AZD5004(Part B) — AZD5004 will be administered as an oral tablet once daily.
  Arms: Part B-AZD5004
Drug: Placebo(Part B) — Placebo will be administered as an oral tablet once daily.
  Arms: Part B-Placebo

SUMMARY:
This Phase I study will gather important information on the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD5004 in both healthy Japanese participants and Japanese participants with T2DM.

DETAILED DESCRIPTION:
This is a placebo-controlled study to assess the safety, efficacy, tolerability, and PK of single and repeated dosing of AZD5004 compared with placebo.

Participants who are eligible according to the inclusion/exclusion criteria will be randomized to receive AZD5004 or matching placebo.

The study will comprise:

1. A Screening Period of maximum 28 days.
2. A Treatment Period of 1 day(Part A) or 105 days (Part B).
3. A final Follow-up Visit approximately 7 days(Part A) or 14 days(Part B) after the last study intervention administration.

ELIGIBILITY:
Inclusion Criteria:

* Japanese men or women, and 18-65 years of age inclusive, at the time of signing the informed consent.

Inclusion Criteria for Part A:

* HbA1c ≤ 6.0%.
* Body weight ≥ 50.0 kg and BMI within the range 18.0-32.0 kg/m2.

Inclusion Criteria for Part B:

* HbA1c ≥ 6.5% and ≤ 10.5%.
* Not on any other diabetic medications.
* Body weight ≥ 60.0 kg and BMI within the range 24.0-35.0 kg/m2

Exclusion Criteria:

* Has a clinically relevant acute or chronic medical condition or disease.
* History of acute pancreatitis and chronic pancreatitis, gallstones.
* Abnormal renal function.
* Known clinically significant gastric emptying abnormality
* Significant hepatic disease.
* Uncontrolled thyroid disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
PartA: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28) to last follow up visit (Day 8)
  To assess the safety and tolerability of AZD5004 following single oral doses in healthy participants.
PartB: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28) to last follow up visit (Day 119 )
  To assess the safety and tolerability of AZD5004 following multiple oral ascending doses in participants with T2DM.

SECONDARY OUTCOMES:
PartB: AUC0-4 for glucose, insulin and C-peptide for MMTT | From Day 1 to Day 105
  To describe the PD of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Absolute change from baseline to Day 105 in fasting plasma glucose | From Day 1 to Day 105
  To describe the PD of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: % change from baseline to Day 105 in HOMA-IR | From Day 1 to Day 105
  To describe the PD of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: The proportion of time in hyperglycaemia /hypoglycaemia over the last 7-day intervals at each dose level in CGM | From Day 1 to Day 106
  To describe the PD of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: % change from baseline to Day 105 in body weight (kg) | From Day 1 to Day 105
  To describe the PD of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: % change from baseline to Day 105 in waist circumference (cm) | From Day 1 to Day 105
  To describe the PD of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartA: Area under the Plasma Concentration vs. Time Curve(AUC0-24) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Area under the Plasma Concentration vs. Time Curve from Zero until the Time of the Last Concentration above the Limit of Quantification(AUC0-tlast) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Area under the Plasma Concentration vs. Time Curve from Zero to Infinity(AUC0-inf) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Maximum Observed Plasma Concentration(Cmax) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Plasma Concentration at 24 Hours Post-Dose(C24h) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Time of Occurrence of Maximum Plasma Concentration(tmax) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Lag Time before Observation of Quantifiable Analyte Concentrations in Plasma(tlag) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Half-Life(t1/2) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Last measurable Non-Zero Concentration(Clast) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Last measurable Non-Zero ConcentrationTime to Last Detectable Concentration(tlast) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Apparent Oral Clearance(CL/F) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Cumulative Urinary Excretion(Ae) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartA: Clearance(CLR) | From Day 1 to Day 6
  To describe the PK (plasma and urine) of AZD5004 following a single administration in healthy participants in SAD
PartB: Area under the Plasma Concentration vs. Time Curve(AUC0-24) | Day 1
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Maximum Observed Plasma Concentration(Cmax) | Day 1, Day 49, Day 63, Day 77, Day91, Day105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Plasma Concentration at 24 Hours Post-Dose(C24h) | Day 1
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Time of Occurrence of Maximum Plasma Concentration(tmax) | Day 1, Day 49, Day 63, Day 77, Day91, Day105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Lag Time before Observation of Quantifiable Analyte Concentrations in Plasma(tlag) | Day 1
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Area under the Plasma Concentration vs. Time Curve over the Dosing Interval(AUC0-τ) | Day 49, Day 63, Day 77, Day 91, Day 105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Observed Concentration at the End of the Dosing Interval(Cτ) | Day 49, Day 63, Day 77, Day 91, Day 105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Half-Life(t1/2) | Day 49, Day 63, Day 77, Day 91, Day 105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Apparent Oral Clearance(CL/F) | Day 49, Day 63, Day 77, Day 91, Day 105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Cumulative Urinary Excretion(Ae) | Day 105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD
PartB: Clearance(CLR) | Day 105
  To describe the PK (plasma and urine) of AZD5004 following repeated daily administration in participants with T2DM in MAD

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/